CLINICAL TRIAL: NCT04843020
Title: An Open-Label Study of ION-682884 in Patients With TTR Amyloidosis Who Have Completed a 24-Open Label Study of Inotersen for TTR Amyloidosis Cardiomyopathy
Brief Title: ION-682884 in Patients With TTR Amyloid Cardiomyopathy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Rodney H. Falk, MD, Director, BWH Amyloidosis Program, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021P000784
Record Dates: First submitted 2021-04-05; First posted 2021-04-13 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Transthyretin Amyloid Cardiopathy
Keywords: amyloidosis; transthyretin; antisense oligonucleotide; ION682884; cardiomyopathy
MeSH Terms: conditions — Amyloidosis; Cardiomyopathies

STUDY DESIGN:
Intervention Model Description: open label study of investigational antisense oligonucleotide targeting TTR
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Drug subcutaneous injection (Experimental): Monthly injection of ION 682884, administered subcutaneously at a dose of 45 mg.
  Interventions: Drug: ION 682884

INTERVENTIONS:
Drug: ION 682884 — Subcutaneous injection every month

SUMMARY:
Transthyretin is a protein produced in the liver that transports thyroid hormone and vitamin A. A single substitution of an amino acid in the structure of TTR can result in a relatively unstable protein, the breakdown products of which (predominantly monomers) aggregate abnormally and produce proteinaceous deposits in nerves and the heart. These deposits are known as amyloid and produce progressive nerve and heart damage. Amyloidosis due to a mutant TTR is usually an autosomal dominant and hence is a familial condition. Wild-type TTR is also capable of producing amyloid deposits which predominantly involves the heart (rather than the nervous system) resulting in a progressive decrease in cardiac function with increasing signs of heart failure. This study aims to determine whether subcutaneous injection of an antisense oligonucleotide drug, known as ION-682884, that has been specifically designed to reduce production of the protein transthyretin by the liver, can slow or stop the progression of TTR amyloid cardiomyopathy as compared to historical controls, using advanced echocardiography and cardiac MRI. This study drug will only be administered to patients who have completed a 24-month study of a similar drug, inotersen (clinicaltrials.gov identifier NCT037028289).The study also aims to determine the tolerability and safety of this drug when administered over a 36+-month period to patients with TTR amyloid cardiomyopathy. The study duration is open-ended and will continue either until this agent is approved by the FDA, or production is discontinued based on results of ongoing double-blinded studies.

DETAILED DESCRIPTION:
The study is limited to those patients who have completed 24 months in our single-center open-label trial of inotersen for amyloid cardiomyopathy (NCT037028289). Patients must have an estimated glomerular filtration rate of greater than 30 and a platelet count greater than 130,000. They will have either wildtype or mutant transthyretin cardiomyopathy. It is anticipated that up to 17 patients will be eligible for the study, age 65-85 years.

Research design:

After completion of the 24 months in the inotersen study, patients will undergo their final visit and assessment. This will include an echocardiogram, lab work, 6-minute walk test, cardiopulmonary exercise testing and, in those without a pacemaker, a cardiac MRI. If the lab work from the end of study confirms eligibility for the new study, patients will be offered the option of continuing with the TTR-lowering drug, ION-682884. After informed consent the patient will be supplied with prefilled syringes containing ION-682884 and the first injection administered. They will return for follow up visits at six weeks, 12 weeks, three months, and six months thereafter. At each six-monthly visit they will undergo the same testing as they had in the inotersen study, namely laboratory measurements, 6-minute walk test, cardiopulmonary exercise testing, echocardiogram and, unless contraindicated, cardiac MRI. The patients will remain in the study for an open-ended period of time until study ending criteria occur (reduction in the glomerular filtration rate to less than 30 or platelet count with a significant fall) or until the drug is FDA-approved or the manufacturer or principal investigator terminates the study.

Because ION-682884 is an antisense oligonucleotide similar to inotersen and because inotersen has been associated with thrombocytopenia and worsening renal function, patients will have weekly lab draws done in their own home for safety monitoring. These bloods will be used to measure platelet function every week, and renal function every other week. This is currently mandated by the Food and Drug administration in the double-blinded study of ION-682884 but the frequency of blood draws may be decreased overtime depending on the interim safety analysis results from that study and FDA evaluation of that data.

ELIGIBILITY:
Inclusion Criteria:

1. Only patient who have completed 24 months of therapy in the open label clinical trial of inotersen, "A 24-month open-label study of the tolerability and efficacy of an antisense oligonucleotide (inotersen) in patients with transthyretin (TTR) amyloid cardiomyopathy" (Protocol #:2018-P001436) will be enrolled. All patients in that study had either wild-type transthyretin amyloidosis (ATTRwt) or mutant transthyretin amyloidosis (ATTRm) cardiac amyloidosis, defined by standard criteria. Additional criteria for the current study are as follows:

1. Patients should, in the opinion of the Investigator, be in a stable state in terms of New York Heart Association (NYHA) class. Class I-III patients will be recruited.
2. Age 65-85 years
3. Male, or non-pregnant, non-lactating females. If a male partners with a premenopausal woman, he must be willing to use the following methods of contraception: condoms, oral/hormonal contraception, Intrauterine Device, diaphragm, or abstinence (all patients are either male of post-menopausal) (NB: There will be no premenopausal women in the proposed study)
4. Written informed consent to be obtained prior to study treatment
5. Willingness to return to the treating center for follow-up
6. Willingness and ability to self-administer, or to have spouse administer subcutaneous injections of study drug every 4 weeks.
7. Willingness to take oral Vitamin A supplementation throughout the study and for 3 months thereafter.

Exclusion Criteria:

1. Acute coronary syndrome, unstable angina, stroke, transient ischemic attack,, coronary revascularization, cardiac device implantation, cardiac valve repair, or major surgery within 3 emergency room for worsening of HF with discharge date within 4 weeks prior to or during Screening 3. Uncontrolled hypertension (systolic blood pressure [BP] > 160 or diastolic BP > 100 mmHg) 4. Uncontrolled clinically significant cardiac arrhythmia, per Investigator's assessment (e.g., no pacemaker, although indicated) 5. Severe uncorrected cardiac valvular disease 6. Cardiomyopathy not primarily caused by amyloidosis, for example, cardiomyopathy due to hypertension, valvular heart disease, or ischemic heart disease 7. Screening laboratory results as follows, or any other clinically significant abnormalities in Screening laboratory values that would render a patient unsuitable for inclusion

1. Alanine aminotransferase/aspartate aminotransferase (ALT/AST) > 2.0 × upper limit of normal (ULN)
2. Total bilirubin ≥ 1.5 × ULN (patients with total bilirubin ≥ 1.5 × ULN may be allowed on study if indirect bilirubin only is elevated, ALT/AST is not greater than the ULN and known to have Gilbert's disease)
3. Platelets < 125 × 109/L
4. Urine protein creatinine ratio (UPCR) ≥ 750 mg/g. In the event of UPCR above this threshold ineligibility may be confirmed by a repeat random spot UPCR ≥ 750 mg/g
5. Positive test for blood (including trace) on urinalysis that is subsequently confirmed with urine microscopy showing > 5 red blood cells per high power field and is related to glomerulopathies. In women, this exclusion criterion must be assessed outside of menstrual period. If in the opinion of the Investigator the hematuria is not considered related to glomerulopathies the patient may be considered eligible, pending proper follow-up and a discussion with the Medical Monitor. Patients with history of bladder cancer must have been treated with curative intent and have not presented recurrence within the prior 5 years
6. Estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m2 at Screening. If the eGFR is thought to be underestimated, the CKD-EPI creatinine-cystatin C equation can be used for confirmation.
7. Abnormal thyroid function tests with clinical significance per Investigator judgement
8. Hemoglobin A1c (HbA1c) > 9.5% 8. Monoclonal gammopathy of undetermined significance (MGUS) and/or alterations in immunoglobulin free light chain (FLC) ratio, unless fat, bone marrow, or heart biopsy confirming the absence of light chain and the presence of TTR protein by mass spectrometry or immunoelectron microscopy. For patients with CKD and without presence of monoclonal protein in blood and urine, the acceptable FLC ratio is 0.26-2.25.

   9. Active infection requiring systemic antiviral or antimicrobial therapy that will not be completed prior to Study Day 1 10. Known history of or positive test for human immunodeficiency virus (HIV) (as evidenced by positive tests for HIV antibody and HIV RNA), hepatitis C (as evidenced by positive tests for HCV antibody and HCV RNA) or hepatitis B (as evidenced by a positive test for hepatitis B surface antigen) 11. History of bleeding, diathesis or coagulopathy (e.g., liver cirrhosis, hematologic malignancy, antiphospholipid antibody syndrome, congenital disorders such as hemophilia A, B, and Von Willebrand disease) 12. If receiving oral anticoagulants (except vitamin K antagonists), the dose must have been stable for 4 weeks prior to the first dose of Study Drug and regular monitoring must be performed, per clinical practice during the study. If the patient is receiving vitamin K antagonists (e.g., warfarin) INR should be in therapeutic range, as established by the Investigator, for 4 weeks prior to the first dose 13. Malignancy within 5 years, except for basal or squamous cell carcinoma of the skin, melanoma in situ, prostate carcinoma grade group 1, breast ductal carcinoma in situ, or carcinoma in situ of the cervix successfully treated. Patients with a history of other malignancies who have been treated with curative intent and without recurrence within 5 years may also be eligible per Investigator judgment 14. Prior liver or heart transplant, and/or Left Ventricular Assist Device (LVAD) or anticipated liver transplant or LVAD within 1 year after randomization 15. Karnofsky performance status of ≤ 50% 16. Contraindication for immunosuppressive therapy, per Investigator's discretion 17. Known Light chain/Primary Amyloidosis (AL) 18. Known leptomeningeal amyloidos

   -

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Echocardiographic change | 48 months
  change in echocardiographically-derived left ventricular longitudinal strain (measured as percentage change from end diastole to end systole)
Change in cardiac MRI | 48 months
  Change in extracellular volume (measure as a percentage of total of LV mass) between baseline MRI and 48 months
Change in cardiac MRI | 48 months
  Change in left ventricular mass, measured by cardiac MRI (gm/m2) , between baseline and 48 months
change in 6 minute walk | 48 months
  change in distance walked (measured in meters) between baseline 6 minute walk and walk after 48 months of therapy
change in cardiopulmonary testing | 48 months
  change in maximal oxygen consumption (VO2 max measured in ml/kg.min) between baseline cardiopulmonary testing and cardiopulmonary testing at 48 months of therapy
change in the cardiac biomarker NTproBNP | 48 months
  change between baseline and after 48 months of therapy of serum NTproBNP (measured in pg/ml)
change in the cardiac biomarker high-sensitivity troponin | 48 months
  change between baseline and after 48 months of therapy of serum high-sensitivity troponin T measured in ng/L)

SECONDARY OUTCOMES:
Response of transthyretin levels to therapy | 3 months
  Absolute decrease in TTR levels (measured in mg/dl) after initiation of therapy, compared to response, in previous study, to weekly inotersen injections.
Time frame of response of TTR levels to therapy | 3 months
  Time frame to nadir of TTR levels (weeks) after initiation of therapy, compared to response, in previous study, to weekly inotersen injections.
Side-effect profile: renal function | 48 months
  Effect of therapy on renal function, measured as estimated glomerular filtration rate (mL/min/1.73m2), between baseline measurements and 48 months, measured every 2 weeks
Side effect profile: platelets | 48 months
  Effect of therapy on platelet count (normal 150,000 - 450,000/uL), between baseline measurements and 48 months, measured every week

CONTACTS AND LOCATIONS:
Overall Officials: Rodney H Falk, Study Director — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No